CLINICAL TRIAL: NCT06485596
Title: Direct Procurement (DP) and Hypothermic Oxygenated Perfusion (HOPE) of Donor Hearts After Circulatory Death (DCD) Using the XVIVO Heart Assist Transport System
Brief Title: HOPE At Heart (HOPE) of Donor Hearts After Circulatory Death (DCD) Using the XVIVO Heart Assist Transport System.
Acronym: HOPE@Heart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: XVIVO Perfusion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOPE at Heart
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DCD Direct procurement (Experimental): Direct procurement of DCD donor hearts
  Interventions: Device: XVIVO Heart Assist Transport System

INTERVENTIONS:
Device: XVIVO Heart Assist Transport System — Direct procurement of donor hearts from DCD donation
  Other Names: Direct procurement

SUMMARY:
The purpose of the clinical investigation is to support the use of direct procurement of donor hearts in donation after circulatory death followed by hypothermic oxygenated perfusion using the XVIVO Heart Assist Transport System. Thereby increasing the utilization of DCD donor hearts in donation after circulatory death.

The primary objective is to evaluate patient survival after direct procurement and hypothermic oxygenated machine perfusion of DCD donor hearts using the XVIVO Heart Assist Transport System.

The secondary objectives are to evaluate patient outcomes and graft function post-transplant.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-national, multicentre, proof-of-concept study to evaluate post-transplant outcomes after the use of direct procurement followed by a period of hypothermic oxygenated perfusion of the donor heart in DCD using the XVIVO Heart Assist Transport system.

The investigation will be conducted at 4 heart transplant centres, one in Belgium and three in The Netherlands.The study will include 20 DCD heart transplant recipients and will evaluate transplant outcomes such as post-transplant complications, patient survival and graft function for a period of 6 months post-transplant.

The study will not include a control group as this is a proof-of-concept study, investigating an alternative method of procurement of DCD hearts by providing additional safety and performance data.

The primary objective is to evaluate patient survival after direct procurement and hypothermic oxygenated machine perfusion of DCD donor hearts using the XVIVO Heart Assist Transport System.

The secondary objectives are to evaluate patient outcomes and graft function post-transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Signed informed consent form
3. Accepted and/or listed for heart transplantation

Exclusion Criteria:

1. Not able to understand the information provided during the informed consent procedure
2. Previous solid organ transplantation
3. Grown-up congenital heart disease
4. Dialysis
5. Incompatible blood group
6. Combined organ transplantation candidates
7. Subjects under pre-transplant desensitization protocol (including plasma exchange in conjunction with the transplant surgery)
8. Mechanical circulatory support pre-transplantation (except durable Left ventricular assist device or Intra-aortic balloon pump)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Patient survival | 30 days post-transplant

SECONDARY OUTCOMES:
Cardiac related mortality | 30 days post-transplant
Incidence of Mechanical circulatory support | 30 days post-transplant
Incidence of severe Primary Graft Dysfunction (PGD) at 24 hours post-transplant (Kobashigawa et al., 2014) | 30 days post-transplant
Cardiac function as assessed by left ventricular ejection fraction (LVEF) at 24 hours and 30 days post-transplant | 30 days post-transplant
Incidence of perfused hearts which are not used for transplantation | 30 days post-transplant
Total duration of ICU stay (days) | 30 days post-transplant
Incidence of biopsy proven rejections > 1 ACR (leading to changed immunosuppressive regime) | 30 days post-transplant
Cardiac related mortality at 6 months post-transplant | 6 months post-transplant
Cardiac function as assessed by left ventricular ejection fraction (LVEF) | 6 months post-transplant
Number of days until hospital discharge from index procedure | 30 days post-transplant
Incidence of biopsy proven rejections > 1 ACR (leading to changed immunosuppressive regime) | 6 months post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Filip Rega, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No